CLINICAL TRIAL: NCT01942265
Title: A Phase II Randomized, Double-Blinded, Controlled Study in Healthy Adults to Assess the Safety, Reactogenicity, and Immunogenicity of a Monovalent Influenza A/H7N9 Virus Vaccine Administered at Different Dosages Given With and Without AS03 and MF59 Adjuvants
Brief Title: H7N9 Mix and Match With AS03 and MF59 in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13-0033; HHSN272200800004C
Record Dates: First submitted 2013-09-04; First posted 2013-09-13 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2014-09

CONDITIONS: Influenza
Keywords: Influenza, Immunogenicity, Monovalent, A/H7N9, Vaccine, AS03, Adjuvant
MeSH Terms: conditions — Influenza, Human | interventions — MF59 oil emulsion; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (10):
- Group 4 (Experimental): 100 subjects receive 15mcg sanofi A/H7N9 antigen plus GSK AS03 adjuvant on Day 0 and 15mcg sanofi A/H7N9 antigen on Day 21
  Interventions: Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 3 (Experimental): 100 subjects receive 15mcg sanofi A/H7N9 antigen plus GSK AS03 adjuvant on Day 0 and 21
  Interventions: Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 1 (Experimental): 100 subjects receive 3.75mcg sanofi A/H7N9 antigen plus GSK AS03 adjuvant on Day 0 and 21
  Interventions: Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 2 (Experimental): 100 subjects receive 7.5mcg sanofi A/H7N9 antigen plus GSK AS03 adjuvant on Day 0 and 21
  Interventions: Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 5 (Experimental): 100 subjects receive 15mcg sanofi A/H7N9 antigen on Day 0 and 15mcg sanofi A/H7N9 antigen plus GSK AS03 adjuvant on Day 21
  Interventions: Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 9 (Experimental): 100 subjects receive 15mcg sanofi A/H7N9 antigen on Day 0 and 21
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 8 (Experimental): 100 subjects receive 15mcg sanofi A/H7N9 antigen plus NVD MF59 adjuvant on Day 0 and 21
  Interventions: Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 7 (Experimental): 100 subjects receive 15mcg sanofi A/H7N9 antigen plus NVD MF59 adjuvant on Day 0 and 15mcg sanofi A/H7N9 antigen plus GSK AS03 adjuvant on Day 21
  Interventions: Drug: AS03; Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 6 (Experimental): 100 subjects receive 15mcg sanofi A/H7N9 antigen plus GSK AS03 adjuvant on Day 0 and 15mcg sanofi A/H7N9 antigen plus NVD MF59 adjuvant on Day 21
  Interventions: Drug: AS03; Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 10 (Experimental): 100 subjects receive 45 mcg sanofi A/H7N9 antigen on Day 0 and 21
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013

INTERVENTIONS:
Drug: AS03 — Subjects will receive two doses of the A/H7N9 vaccine with or without AS03 delivered intramuscularly 21 days apart.
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7
Drug: MF59 — Subjects will receive two doses of the A/H7N9 vaccine with or without MF59 delivered intramuscularly 21 days apart.
  Arms: Group 6; Group 7; Group 8
Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013 — Subjects will receive two doses of the A/H7N9 vaccine with or without an adjuvant delivered intramuscularly approximately 21 days apart.

SUMMARY:
This Phase II randomized, double-blinded, controlled study in up to 1000 males and non-pregnant females, 19 to 64 years old, inclusive, who are in good health and meet all eligibility criteria is designed to provide data on an A/H7N9 vaccine made with HA antigen derived from the influenza A/Shanghai/2/2013 virus.

DETAILED DESCRIPTION:
This Phase II randomized, double-blinded, controlled study in up to 1000 males and non-pregnant females, 19 to 64 years old, inclusive, who are in good health and meet all eligibility criteria is designed to provide data on an A/H7N9 vaccine made with HA antigen derived from the influenza A/Shanghai/2/2013 virus. The study aims to address several critical questions, including the safety, reactogenicity, and immunogenicity of a monovalent influenza A/H7N9 virus vaccine manufactured by Sanofi Pasteur: 1) two doses administered at different dosages (3.75, 7.5, or 15 mcg of HA/0.5 mL dose) given with AS03 adjuvant manufactured by GlaxoSmithKline Biologicals or without adjuvant (15 mcg of HA/0.5 mL dose and 45 mcg of HA/0.75 mL dose); and 2) a combination of two doses of the A/H7N9 vaccine (15 mcg of HA/0.5 mL dose) each administered with a different adjuvant (AS03 or MF59 manufactured by Novartis Vaccines and Diagnostics); and 3) two doses administered at 15 mcg of HA/0.5 mL dose given with MF59 adjuvant manufactured by Novartis Vaccines and Diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to initiation of any study procedures.
* Are able to understand and comply with planned study procedures and be available for all study visits.
* Are males or non-pregnant females, 19 to 64 years old, inclusive.
* Are in good health, as determined by vital signs (oral temperature, pulse, and blood pressure), medical history, and targeted physical examination based on medical history to ensure any existing medical diagnoses or conditions (except those in the Subject Exclusion Criteria) are stable . Subjects may be on chronic1 or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity. Note: Topical, nasal, and inhaled medications (with the exception of steroids as outlined in the Subjects Exclusion Criteria (see Section 5.2), vitamins, and contraceptives are permitted.
* Oral temperature is less than 100.4 degrees F.
* Pulse is 50 to 115 bpm, inclusive.
* Systolic blood pressure is 85 to 150 mm Hg, inclusive.
* Diastolic blood pressure is 55 to 95 mmHg, inclusive.
* Erythrocyte sedimentation rate (ESR) is less than 30 mm per hour.
* Alanine aminotransferase (ALT) is less than 44 IU/L for females or is less than 61 IU/L for males.
* Creatinine is less than 1.11 mg/dL for females or is less than 1.38 mg/dL for males.
* White blood cells (WBC) are greater than 3.9 x10^3/UL and less than 10.6 x10^3/UL.
* Hemoglobin is greater than 11.4 g/dL for females or is greater than 12.4 g/dL for males.
* Platelets are greater than 139 x10^3/UL and less than 416 x10^3/UL.
* Total bilirubin is less than 1.3 mg/dL.
* Female subjects of childbearing potential who are not surgically sterile via tubal sterilization, bilateral oophorectomy, or hysterectomy or who are not postmenopausal for >/= 1 year must agree to practice highly effective contraception that may include, but is not limited to, abstinence from intercourse with a male partner, monogamous relationship with a vasectomized partner, male condoms with the use of applied spermicide, intrauterine devices, and licensed hormonal methods with use of a highly effective method of contraception for a minimum of 30 days prior to study product exposure and agree to practice highly effective contraception for the duration of study product exposure, including 2 months (defined as 60 days) after the last study vaccination. A highly effective method of contraception is defined as one which results in a low failure rate (i.e., less than 1 percent per year) when used consistently and correctly. Method of contraception will be captured on the appropriate data collection form.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

* Have an acute illness within 72 hours prior to study vaccination.
* Have any condition that, in the opinion of the site principal investigator or appropriate sub-investigator, would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or confound the interpretation of the results.
* Have an acute or chronic medical condition that, in the opinion of the site principal investigator or appropriate sub-investigator, would render vaccination unsafe, or would interfere with the evaluation of responses.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
* Have known active neoplastic disease or a history of any hematologic malignancy.
* Have known HIV, hepatitis B, or hepatitis C infection.
* Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.
* Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
* Have a personal or family history of narcolepsy with or without cataplexy.
* Have a history of Guillain-Barré Syndrome.
* Have a history of neuralgia, paresthesia, neuritis, convulsions, or encephalomyelitis within 90 days prior to study vaccination.
* Have a history of autoimmune disease, including but not limited to neuroinflammatory diseases, vasculitis, clotting disorders, dermatitis, arthritis, thyroiditis, or muscle, liver or kidney disease.
* Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
* Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
* Have taken oral or parenteral corticosteroids of any dose within 30 days prior to study vaccination.
* Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination. High-dose defined as >800mcg/day of beclomethasone dipropionate CFC or equivalent.
* Received any licensed live vaccine within 30 days or any licensed inactivated vaccine within 14 days prior to the first study vaccination or planned receipt of any vaccine from the first study vaccination through the follow-up visit at approximately 21 days after the last study vaccination. This is inclusive of licensed seasonal influenza vaccines.
* Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 30 days prior to the first study vaccination, or expects to receive an experimental agent other than from participation in this study during the 13-month study period.
* Are participating or plan to participate in another clinical trial with an interventional agent (licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) during the 13-month study period.
* Prior participation in a clinical trial of influenza A/H7 vaccine and assigned to a group receiving influenza A/H7 vaccine (does not apply to documented placebo recipients) or have a history of A/H7 actual or potential exposure or infection prior to the first study vaccination.
* Plan to travel outside the U.S. (continental U.S., Hawaii and Alaska) in the time between the first study vaccination and 42 days after the first study vaccination.
* Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after their last study vaccination.
* Blood donation within 30 days prior to enrollment and within 30 days after the last blood draw (only for a subset of healthy adult subjects - all volunteers, 19-64 years old, enrolled at the Vanderbilt VTEU site, who consent to blood donation for the immunology exploratory assays).

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 980 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving seroconversion (defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer >/=1:40 or a pre-vaccination HAI titer >/=1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer). | Day 42 (21 days post second study vaccination)
Occurrence of solicited injection site and systemic reactogenicity on the day of each study vaccination through 7 days after each study vaccination. | Day 0 though Day 29
Occurrence of study vaccine-related serious adverse events from the time of the first study vaccination through approximately 13 months after the first study vaccination. | Day 0 through Day 386
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the study vaccine at approximately 21 days after the second study vaccination. | Day 42 (21 days post second study vaccination)
Occurrence of clinical safety laboratory adverse events from the time of each study vaccination through approximately 8 days after each study vaccination. | Day 0 through Day 29

SECONDARY OUTCOMES:
Percentage of subjects achieving seroconversion (defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer >/=1:40 or a pre-vaccination HAI titer >/=1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer) | Day 0, 8 and 21
Percentage of subjects achieving seroconversion (defined as either a pre-vaccination Neut titer <1:10 and a post-vaccination Neut titer >/= 1:40 or a pre-vaccination Neut titer >/=1:10 and a minimum four-fold rise in post-vaccination Neut antibody titer) | Day 0, 8, 21, 29, and 42
Percentage of subjects achieving seroconversion (defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer >/=1:40 or a pre-vaccination HAI titer >/=1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer). | Day 29 (8 days after the second study vaccination)
Occurrence of unsolicited adverse events from the time of the first study vaccination through approximately 21 days after the last study vaccination. | Day 42 (21 days post last study vaccination
Geometric Mean Titers of serum HAI and Neut antibody at baseline and at approximately 8 and 21 days after each study vaccination. | Days 0, 8, 21, 29, and 42
Percentage of subjects achieving a serum Neut antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the study vaccine at baseline and at approximately 8 and 21 days after each study vaccination | Day 0, 8, 21, 29, and 42
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the study vaccine at approximately 8 days after the second study vaccination. | Day 29 (8 days after the second study vaccination)
Occurrence of new-onset chronic medical conditions through 13 months after the first study vaccination. | Through Day 386 (13 months after the first vaccination)
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the study vaccine at baseline and at approximately 8 and 21 days after the first study vaccination. | Days 0, 8 and 21

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Vanderbilt University Medical Center - Infectious Diseases, Nashville, Tennessee
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle - Vaccines and Infectious Diseases, Seattle, Washington

REFERENCES:
- [Result] Jackson LA, Campbell JD, Frey SE, Edwards KM, Keitel WA, Kotloff KL, Berry AA, Graham I, Atmar RL, Creech CB, Thomsen IP, Patel SM, Gutierrez AF, Anderson EL, El Sahly HM, Hill H, Noah DL, Bellamy AR. Effect of Varying Doses of a Monovalent H7N9 Influenza Vaccine With and Without AS03 and MF59 Adjuvants on Immune Response: A Randomized Clinical Trial. JAMA. 2015 Jul 21;314(3):237-46. doi: 10.1001/jama.2015.7916. PMID 26197184